CLINICAL TRIAL: NCT02161770
Title: An Open-label, Non-randomised, Multicentre, Comparative, Phase I Study to Determine the Pharmacokinetics, Safety and Tolerability of AZD9291 Following a Single Oral Dose to Patients With Advanced Solid Tumours and Normal Hepatic Function or Mild or Moderate Hepatic Impairment
Brief Title: Study to Assess the Blood Levels and Safety of AZD9291 in Patients With Advanced Solid Tumours and Normal Liver Function or Mild or Moderate Liver Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D5160C00008; 2014-001515-39 (EudraCT Number)
Record Dates: First submitted 2014-05-29; First posted 2014-06-12 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Solid Tumours
Keywords: oncology, cancer, neoplasm, anticancer drug, pharmacokinetics, area under curve, AZD9291, solid tumour, mild hepatic impairment, moderate hepatic impairment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal hepatic function (Other): Patients without a history or presence of hepatic disease
  Interventions: Drug: AZD9291 tablet dosing; Procedure: Pharmacokinetic sampling - AZD9291; Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550
- Mild hepatic impairment (Other): Patients defined by the Child-Pugh classification system to be Child-Pugh A
  Interventions: Drug: AZD9291 tablet dosing; Procedure: Pharmacokinetic sampling - AZD9291; Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550
- Moderate hepatic impairment (Other): Patients defined by the Child-Pugh classification system to be Child-Pugh B
  Interventions: Drug: AZD9291 tablet dosing; Procedure: Pharmacokinetic sampling - AZD9291; Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550

INTERVENTIONS:
Drug: AZD9291 tablet dosing — Part A - single 80mg oral dose AZD9291 (administered as 1 80mg tablet). Part B - 80mg oral dose AZD9291 od.
Procedure: Pharmacokinetic sampling - AZD9291 — Blood sampling to measure AZD9291 pharmacokinetic parameters.
Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550 — Blood samples to measure the pharmacokinetic parameters of AZ5104 and AZ7550.

SUMMARY:
This is a 2-part study in patients with advanced solid tumours. Part A will investigate the pharmacokinetics (PK) of AZD9291 in patients with mild or moderate hepatic impairment compared to patients with normal hepatic function; Part B will allow any patient with mild or moderate hepatic impairment or normal hepatic function, who completes Part A, continued access to AZD9291 after the PK phase and will provide additional safety data.

ELIGIBILITY:
For inclusion in the study as a patient with hepatic impairment, the following criterion must be met:

1. Patients must have stable chronic hepatic impairment for at least 2 weeks prior to Day 1, see Section 4.1.1. Patients with hepatic metastases and/or HCC are eligible for the study, providing the hepatic metastases or HCC are not the sole reason for any changes in liver function satisfying the criteria for mild or moderate hepatic impairment as defined by the Child Pugh criteria. Patients must have globally impaired hepatic function to participate in the study.

For inclusion in the study as a patient with normal hepatic function, the following criteria must be met:

1. Negative result for serum hepatitis B surface antigen and hepatitis C antibody
2. Total bilirubin less than or equal to1.5 x institutional ULN, albumin and prothrombin time within normal limits and must not have ascites (unless related to disease under study) or encephalopathy.
3. AST and ALT less than or equal to2.5 x institutional ULN unless liver metastases are present in which case it must be less than or equal to5 x ULN.

All patients must fulfil the following criteria:

1. Male or female, aged at least 18 years.
2. Histological or, where appropriate, cytological confirmation of any malignant solid tumour refractory or resistant to standard therapy or for which no suitable effective standard therapy exists. Tumours in which inhibition of the EGFR pathway is considered relevant by the Investigator are not mandated but are encouraged.
3. ECOG performance status less than or equal to2.
4. Patients must have a life expectancy of greater than or equal to12 weeks, as estimated at the time of screening.
5. Females should be using adequate contraceptive measures and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening: post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments; women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the postmenopausal range for the institution; documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
6. Male patients should be willing to use barrier contraception, ie, condoms, until 6 months after last study drug is taken.

Exclusion criteria:

1. Participation in another clinical study with an IP during the last 14 days (or a longer period depending on the defined characteristics of the agents used).
2. Treatment in the previous 3 months before dosing in this study with any drug known to have a well-defined potential for fulminant hepatotoxicity (eg, halothane and methotrexate).
3. Treatment with any of the following: an EGFR TKI w/in 8 days or approximately 5x half-life, whichever is the longer, of the first dose of study treatment; Any cytotoxic chemotherapy, investigational agents or other anticancer drugs w/in 14 days of the first dose of study treatment; Major surgery (excluding placement of vascular access) w/in 4 weeks of the first dose; Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within 4 weeks of the first dose of study treatment; Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inhibitors of CYP3A4 (at least 1 week prior) and potent inducers of CYP3A4 (at least 3 week prior) (Appendix H). All patients in Part B and continued access must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known potent inducer/inhibitory effects on CYP3A4 (Appendix H).
4. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2 prior platinum-therapy related neuropathy.
5. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of the IP until final PK sample collection on Day 22.
6. Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to start of study treatment.
7. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
8. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values: ANCless than1.5x10.9/L; platelet count less than100x10.9/L; haemoglobinless than90 g/L; Creatinine greater than1.5 x institutional ULN concurrent with creatinine clearance less than50 mL/min (measured or calculated by Cockcroft-Gault formula); confirmation of creatinine clearance is only required when creatinine is greater than1.5 x institutional ULN.
9. Any of the following cardiac criteria: Mean resting corrected QT interval corrected for heart rate using Fridericia's correction factor (QTcF) greater than470 msec obtained from 3 ECGs; Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block, second degree heart block, PR interval greater than250 msec; Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval.
10. Patients unable to swallow oral medication or patients with GI disorders or significant GI resection likely to interfere with the absorption of AZD9291.
11. Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
12. Women who are breastfeeding.
13. Patients with a known hypersensitivity to AZD9291 or any of its excipients. Patients with normal hepatic function should not have a history or presence of hepatic disease known to interfere with the absorption, distribution, metabolism or excretion of AZD9291.

Patients with mild or moderate hepatic function should not enter if the following are fulfilled:

1. Patients with hepatic encephalopathy within the last 4 weeks prior to Day 1.
2. Fluctuating or rapidly deteriorating hepatic function as indicated by widely varying or worsening of clinical and/or laboratory signs of hepatic impairment within the screening period.
3. Presence of acute liver disease caused by drug toxicity or by an infection.
4. Severe portal hypertension or surgical porto-systemic shunts.
5. Biliary obstruction or other causes of hepatic impairment not related to parenchymal disorder and/or disease of the liver.
6. Oesophageal variceal bleeding within the past 2 months.
7. Anticoagulant therapy with warfarin or related coumadine.NOTE: Preferred format includes lists of inclusion and exclusion criteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12-22 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of AZD9291 by assessment of maximum plasma AZD9291 concentration (Cmax) | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Rate and extent of absorption of AZD9291 following single oral doses of AZD9291 tablet formulation by assessment of maximum plasma AZD9291 concentration (Cmax).
Pharmacokinetics of AZD9291 by assessment of area under the plasma concentration time curve from zero to infinity (AUC) | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Rate and extent of absorption of AZD9291 following single oral doses of AZD9291 tablet formulation by assessment of area under the plasma concentration time curve from zero to infinity (AUC).

SECONDARY OUTCOMES:
Pharmacokinetics of AZD9291, AZ5104, and AZ7550 by assessment of AUC(0-t) | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Rate and extent of absorption of AZD9291 by assessment of AUC from time zero to last quantifiable dose AUC(0-t)
Pharmacokinetics of AZ5104 and AZ7550 by assessment of Cmax | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Assessment of the PK of AZ5104 and AZ7550 using maximum plasma concentration (Cmax).
Assessment of the safety and tolerability of AZD9291 | Parts A and B, approximately seven months
  Safety data collected using: Assessment of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v4.0; Vital signs (blood pressure, pulse, temperature, height, weight); laboratory parameters (clinical chemistry, haematology, urinalysis); physical examination; and standard 12-lead electrocardiograms (ECGs)
Pharmacokinetics of AZD9291, AZ5104, and AZ7550 by assessment of tmax | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Rate and extent of absorption of AZD9291, AZ5104, and AZ7550 by assessment of time to Cmax (tmax)
Pharmacokinetics of AZD9291, AZ5104, and AZ7550 by assessment of AUC(0-24) | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Rate and extent of absorption of AZD9291, AZ5104, and AZ7550 by assessment of AUC from time zero to t=24, AUC(0-24)
Pharmacokinetics of AZD9291, AZ5104, and AZ7550 by assessment of AUC(0-72) | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Rate and extent of absorption of AZD9291, AZ5104, and AZ7550 by assessment of AUC from time zero to t=72, AUC(0-72)
Pharmacokinetics of AZD9291, AZ5104, and AZ7550 by assessment of AUC(0-168) | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Rate and extent of absorption of AZD9291, AZ5104, and AZ7550 by assessment of AUC from time zero to t=168, AUC(0-168).
Pharmacokinetics of AZD9291, AZ5104, and AZ7550 by assessment of λz | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Rate and extent of absorption of AZD9291, AZ5104, and AZ7550 by assessment of terminal rate constant (λz).
Pharmacokinetics of AZD9291, AZ5104, and AZ7550 by assessment of t½ | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Rate and extent of absorption of AZD9291, AZ5104, and AZ7550 by assessment of the terminal half-life (t1/2).
Pharmacokinetics of AZD9291, AZ5104, and AZ7550 by assessment of CL(R) | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Rate and extent of absorption of AZD9291, AZ5104, and AZ7550 by assessment of renal clearance (CL(R).
Pharmacokinetics of AZD9291 by assessment of CL/F | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Rate and extent of absorption of AZD9291 by assessment of the apparent clearance following oral administration (CL/F)
Pharmacokinetics of AZD9291 by assessment of Vz/F | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Rate and extent of absorption of AZD9291 by assessment of the apparent volume of distribution (Vz/F)
Pharmacokinetics of AZ5104 and AZ7550 by assessment of AUC | Blood samples are collected at the following timepoints post AZD9291 dose on Day 1: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours
  Assessment of the PK of AZ5104 and AZ7550 using area under the plasma concentration curve from zero extrapolated to infinity (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Rukazenkov, Study Chair — AstraZeneca
Locations (16):
- United States (5):
  - Research Site, San Diego, California
  - Research Site, Atlanta, Georgia
  - Research Site, Detroit, Michigan
  - Research Site, Cleveland, Ohio
  - Research Site, San Antonio, Texas
- Belgium (2):
  - Research Site, Ghent
  - Research Site, Woluwé-St-Lambert
- France (6):
  - Research Site, Angers
  - Research Site, Marseille
  - Research Site, Pierre-Bénite
  - Research Site, Rennes
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
- Research Site, Seoul, South Korea
- Research Site, Madrid, Spain
- Research Site, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Grande E, Harvey RD, You B, Batlle JF, Galbraith H, Sarantopoulos J, Ramalingam SS, Mann H, So K, Johnson M, Vishwanathan K. Pharmacokinetic Study of Osimertinib in Cancer Patients with Mild or Moderate Hepatic Impairment. J Pharmacol Exp Ther. 2019 May;369(2):291-299. doi: 10.1124/jpet.118.255919. Epub 2019 Mar 14. PMID 30872388